CLINICAL TRIAL: NCT01940276
Title: A Phase II Open-label, Parallel Group Study of Abiraterone Acetate Plus Prednisone in African American and Caucasian Men With Metastatic Castrate-resistant Prostate Cancer
Brief Title: Abiraterone Race in Metastatic Castrate-resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00046383; 212082PCR2018 (Other: Janssen)
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Results first posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; metastatic; castrate resistant; abiraterone acetate; prednisone; metastatic prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abiraterone Acetate and Prednisone (Experimental): abiraterone acetate will be administered by the patient at a dose of 1000mg orally once daily with prednisone 5 mg BID in 4-week cycles
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone acetate
  Other Names: Zytiga
Drug: Prednisone

SUMMARY:
The primary goal is to prospectively estimate the median radiographic PFS of African American and Caucasian men with mCRPC to abiraterone acetate and prednisone.

DETAILED DESCRIPTION:
This is a non-comparative pilot open-label, parallel arm, multicenter study of abiraterone acetate in African American and Caucasian men with mCRPC. Patients will self-report on race and 50 patients will be enrolled into each group. Patients will be treated on open-label treatment until evidence of disease progression as defined by Prostate Cancer Working Group Two (PCWG2) definition or until two years at which point they will roll over to the standard of care at that time. The study agent abiraterone acetate will be administered by the patient at a dose of 1000mg orally once daily with prednisone 5 mg BID in 4-week cycles throughout the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male, age ≥ 18 years
* Karnofsky performance status ≥ 70
* Life expectancy of ≥ 12 months
* Willing to take abiraterone acetate on an empty stomach; no food should be consumed at least two hours before and for at least one hour after the dose of abiraterone acetate is taken, and should be able to swallow tablets whole, without crushing/chewing tablets
* Patients who have partners of childbearing potential must be willing to use a method of birth control with adequate barrier protection as determined to be acceptable by the principal investigator and sponsor during the study and for 1 week after last dose of abiraterone acetate
* Adequate laboratory parameters
* Histologically confirmed diagnosis of adenocarcinoma of the prostate. Histologic variants of prostate cancer, including neuroendocrine features and small cell carcinoma of the prostate are excluded
* Radiographic evidence of metastatic disease; evaluable non-target lesions and/or bone only metastasis are permitted
* Ongoing ADT using an LHRH agonist (e.g. leuprolide, goserelin) or antagonist (e.g. degarelix) must continue on therapy unless prior bilateral orchiectomy has been performed. Screening serum testosterone must be <50 ng/dl
* PSA ≥ 2.0 ng/mL
* Evidence of of castration resistant disease on ADT as evidenced by one of the following:

  * Absolute rise in PSA of 2.0 ng/mL or greater, minimum 2 consecutive rising PSA levels with an interval of ≥ 1 week between each PSA level, OR
  * 2 consecutive PSA levels 50% or greater above the PSA nadir achieved on ADT and separated at least 1 week apart, OR
  * CT or MRI based evidence of disease progression (soft tissue, nodal or visceral disease progression) according to modified PCWG2 criteria or modified RECIST 1.1 criteria, or at least 1 new bone scan lesion as compared to the most immediate prior radiologic studies)
* A minimum of 2 weeks elapsed off of antiandrogen therapy prior to start of study drug (i.e. flutamide, nilutamide, bicalutamide)
* A minimum of 4 weeks elapsed off of sipuleucel-T prior to start of study drug
* A minimum of 4 weeks from any major surgery prior to start of study drug
* Self-reported race of either African American or Caucasian
* Ability to swallow, retain, and absorb oral medication

Exclusion Criteria:

* Prior treatment with abiraterone acetate or enzalutamide
* Active infection or other medical condition that would make prednisone/prednisolone (corticosteroid) use contraindicated
* Any chronic medical condition requiring a higher dose of corticosteroid than 5mg prednisone/prednisolone bid
* Have known allergies, hypersensitivity, or intolerance to abiraterone acetate or prednisone or their excipients
* Pathological finding consistent with small cell carcinoma of the prostate
* Symptomatic Liver or visceral organ metastasis
* Have a history of gastrointestinal disorders (medical disorders or extensive surgery) that may interfere with the absorption of the study agents
* Known brain metastasis
* Prior cytotoxic chemotherapy or biologic therapy for the treatment of CRPC
* Previously treated with ketoconazole for prostate cancer for greater than 7 days
* Prior systemic treatment with an azole drug (e.g. fluconazole, itraconazole) within 4 weeks of Cycle 1, Day 1
* Uncontrolled hypertension (systolic BP ≥ 160 mmHg or diastolic BP ≥ 95 mmHg). Patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment.
* Poorly controlled diabetes
* Active or symptomatic viral hepatitis or chronic liver disease
* History of pituitary or adrenal dysfunction
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class II-IV heart disease or cardiac ejection fraction measurement of < 50% at baseline
* Atrial Fibrillation or other cardiac arrhythmia requiring therapy
* Other malignancy, except non-melanoma skin cancer, with a ≥ 30% probability of recurrence within 24 months
* Administration of an investigational therapeutic within 30 days of Cycle 1, Day 1
* Any condition which, in the opinion of the investigator, would preclude participation in this trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel George, MD, Principal Investigator — Duke University
Locations (14):
- United States (14):
  - Birmingham VA Medical Center, Birmingham, Alabama
  - Tulane Cancer Center, New Orleans, Louisiana
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Maria Parham Medical Center, Henderson, North Carolina
  - Scotland Memorial Hospital, Laurinburg, North Carolina
  - Southeastern Regional, Lumberton, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - W. G. 'Bill' Hefner VA Medical Center, Salisbury, North Carolina
  - Johnston Memorial Hospital, Smithfield, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Spartanburg Regional, Spartanburg, South Carolina
  - Virginia Oncology Associates, Hampton, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Abiraterone Acetate and Prednisone: White Men: Patients self identifying as white men who received 1000 mg of Abiraterone acetate and 10 mg of prednisone daily till treatment discontinuation.
- Abiraterone Acetate and Prednisone: African American Men: Patients self identifying as African American who received 1000 mg of Abiraterone acetate and 10 mg of prednisone daily till treatment discontinuation.
Period: Overall Study
Arm/Group | Abiraterone Acetate and Prednisone: White Men | Abiraterone Acetate and Prednisone: African American Men
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- White: Patients self identifying as white who received the study regimen
- Black: Patients self identifying as black who received the study regimen
- Total: Total of all reporting groups
Arm/Group | White | Black | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Median (Standard Deviation); unit: years] | 68.2 (7.8) | 69.05 (9.2) | 68.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 50 | 50 | 100
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 50 | 50
  White | 50 | 0 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Median Radiographic Progression Free Survival (PFS)
Description: Time in months from the start of study treatment to the date of first progression according to Prostate Cancer Working Group 2 criteria, or to death due to any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Patients alive who had not progressed as of the last follow-up had PFS censored at the last follow-up date. Median rPFS was estimated using a Kaplan-Meier curve.
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Abiraterone Acetate and Prednisone: White Men: Patients self identifying as white who received 1000 mg of Abiraterone acetate and 10 mg of prednisone daily till treatment discontinuation.
Arm/Group | Abiraterone Acetate and Prednisone: White Men | Abiraterone Acetate and Prednisone: African American Men
Number analyzed (Participants) | 50 | 50
months | 16.8 [11 to 33.7] | 16.6 [12.6 to 22.1]

2. Secondary Outcome: Change in PSA Response
Description: Percent of men with Prostate Specific Antigen (PSA) declines > 30%, > 50% and > 90%
Time Frame: Baseline and up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Abiraterone Acetate and Prednisone: White Men | Abiraterone Acetate and Prednisone: African American Men
Number analyzed (Participants) | 50 | 50
percentage of participants
  Percent of men with PSA declines > 30% | 78 | 82
  Percent of men with PSA declines > 50% | 66 | 74
  Percent of men with PSA declines > 90% | 38 | 48

3. Secondary Outcome: Median Time to PSA Progression
Description: Time to PSA progression as defined by PCWG 2 criteria is the date that a 25% or greater increase and an absolute increase of 2 ng/mL or more from the nadir is documented, which is confirmed by a second value obtained 3 or more weeks later.
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abiraterone Acetate and Prednisone: White Men | Abiraterone Acetate and Prednisone: African American Men
Number analyzed (Participants) | 50 | 50
months | 11.5 [8.5 to 19.3] | 16.6 [11.5 to NA] — Upper limit was not achieved due to insufficient number of participants events

4. Secondary Outcome: Number of Men With PSA Decline to < 0.1 and < 0.2 ng/ml
Description: Number of men who achieve a PSA decline to < 0.1 and < 0.2 ng/ml
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone Acetate and Prednisone: White Men | Abiraterone Acetate and Prednisone: African American Men
Number analyzed (Participants) | 50 | 50
Participants
  PSA decline to < 0.1 | 4 | 9
  PSA decline to < 0.2 | 5 | 13

5. Secondary Outcome: Percent of Subjects Experiencing Hypertension
Description: Incidence and grade of hypertension in the two populations. (Grade 1: Systolic BP 120 to 139 mmHg or diastolic BP 80 to 89 mmHg, Grade 2: Systolic BP 140 to 159 mmHg or diastolic BP 90 to 99 mmHg, Grade 3: Systolic BP ≥160 mmHg or diastolic BP ≥100 mmHg, Grade 4: Life-threatening consequences, urgent intervention indicated)
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone Acetate and Prednisone: White Men | Abiraterone Acetate and Prednisone: African American Men
Number analyzed (Participants) | 50 | 50
Participants
  All grades | 20 | 23
  Grades 3 and 4 | 8 | 12

6. Secondary Outcome: Overall Survival
Description: Length of patient's life after starting study
Time Frame: up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abiraterone Acetate and Prednisone: White Men | Abiraterone Acetate and Prednisone: African American Men
Number analyzed (Participants) | 50 | 50
months | 35.7 [27.1 to NA] — Upper limit was not achieved due to insufficient number of participants events. | 35.9 [24.5 to 43]

ADVERSE EVENTS:
Time Frame: Up to 30 days post last dose
Arm/Group | Abiraterone Acetate and Prednisone: White Men | Abiraterone Acetate and Prednisone: African American Men
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 14/50 | 14/50
Other Adverse Events (participants affected / at risk) | 50/50 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate and Prednisone: White Men (N=50) | Abiraterone Acetate and Prednisone: African American Men (N=50)
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Colonic perforation (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 1 | 1
Pain (General disorders) | 2 | 0
Flu like symptoms (General disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Altered Mental State (Psychiatric disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Squamous cell carcinoma of the face (Skin and subcutaneous tissue disorders) | 1 | 0
Surgical resection of neck cancer (Surgical and medical procedures) | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Acute Congestive Heart Failure (Cardiac disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Accidental Overdose (General disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2
Seizure (Nervous system disorders) | 0 | 1
Transient ischemic attacks (Nervous system disorders) | 0 | 1
Cord Compression (Nervous system disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 2
Hematuria (Renal and urinary disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Asthmatic episode (Respiratory, thoracic and mediastinal disorders) | 0 | 1
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypercapnic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bilaterial pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate and Prednisone: White Men (N=50) | Abiraterone Acetate and Prednisone: African American Men (N=50)
Anemia (Blood and lymphatic system disorders) | 7 | 8
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 2 | 2
White blood cell decreased (Investigations) | 1 | 1
Increased bleeding tendency related to Eliquis (Blood and lymphatic system disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 5 | 5
Alkaline phosphatase increased (Investigations) | 2 | 5
Aspartate aminotransferase increased (Investigations) | 5 | 5
Blood bilirubin increased (Investigations) | 0 | 2
Creatinine increased (Investigations) | 1 | 2
Elevated ANC (Investigations) | 0 | 1
Folic acid deficiency (Investigations) | 1 | 0
Urine output decreased (Investigations) | 0 | 1
Weight gain (Investigations) | 5 | 2
Weight loss (Investigations) | 3 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Acute Congestive Heart Failure (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Irregular heart beat (Cardiac disorders) | 0 | 1
Conduction disorder (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Blurred vision (Eye disorders) | 1 | 1
Dry eye (Eye disorders) | 1 | 0
Conjunctival hemorrhage in right eye (Eye disorders) | 1 | 0
Redness of right eye (Eye disorders) | 0 | 1
Bilateral arcus senilis (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Watering eyes (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Anal hemorrhage (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 14
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 6 | 3
Dry mouth (Gastrointestinal disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 7
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Blood in stool (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 1
Heartburn (Gastrointestinal disorders) | 1 | 0
Hernia (Gastrointestinal disorders) | 1 | 0
Sick (Gastrointestinal disorders) | 0 | 1
Upset stomach (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 8 | 8
Oral pain (Gastrointestinal disorders) | 0 | 2
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 8 | 3
Chills (General disorders) | 0 | 1
Edema face (General disorders) | 0 | 2
Edema limbs (General disorders) | 8 | 13
Fatigue (General disorders) | 21 | 13
Fever (General disorders) | 3 | 2
Flu like symptoms (General disorders) | 5 | 4
Gait disturbance (General disorders) | 1 | 0
Accidental overdose (General disorders) | 0 | 1
Edema face and neck (General disorders) | 0 | 1
Cold-like symptoms (General disorders) | 1 | 0
Overdose (General disorders) | 0 | 1
Irritability (General disorders) | 1 | 0
Localized edema (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2
Pain (General disorders) | 12 | 12
Gallbladder pain (Hepatobiliary disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 2 | 0
Bronchial infection (Infections and infestations) | 3 | 0
Black hairy tongue (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Thrush, related to chemo (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Mouth sores (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 2
Mucosal infection (Infections and infestations) | 0 | 1
Papulopustular rash (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 2 | 4
Urinary tract infection (Infections and infestations) | 5 | 6
Bruising (Injury, poisoning and procedural complications) | 3 | 1
Fall (Injury, poisoning and procedural complications) | 7 | 4
Fracture (Injury, poisoning and procedural complications) | 2 | 1
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 10
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 13
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 2
Hypokalemia (Metabolism and nutrition disorders) | 10 | 17
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 8
Hyponatremia (Metabolism and nutrition disorders) | 2 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 3
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 2
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 3
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1
Back stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Bilateral leg cramps (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasm in right hand (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Bilateral leg weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Bilateral lower leg cramps (Musculoskeletal and connective tissue disorders) | 2 | 0
Burning sensation in bilateral lower extremeties (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 | 1
Right leg aching (Musculoskeletal and connective tissue disorders) | 0 | 1
Weakness, mild and intermittent left upper knee (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 7
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma, neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Smoldering myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 4 | 5
Dysgeusia (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 9 | 3
Memory impairment (Nervous system disorders) | 2 | 1
Movements involuntary (Nervous system disorders) | 1 | 0
Cord Compression (Nervous system disorders) | 0 | 1
Tingling in bilateral legs at HS "like restless legs" (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 5 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 3
Seizure (Nervous system disorders) | 0 | 1
Sinus pain (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient ischemic attacks (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 6
Altered mental state (Psychiatric disorders) | 1 | 0
Altered mental status (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Bladder spasm (Renal and urinary disorders) | 1 | 2
Cystitis noninfective (Renal and urinary disorders) | 2 | 0
Hematuria (Renal and urinary disorders) | 3 | 5
Left hydronephrosis (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 1
Burning during urination (Renal and urinary disorders) | 1 | 0
Burning upon urinating (Renal and urinary disorders) | 0 | 1
Increased BUN (Renal and urinary disorders) | 1 | 0
Pain during urination (Renal and urinary disorders) | 0 | 1
Renal calculi (Renal and urinary disorders) | 2 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 5 | 5
Urinary incontinence (Renal and urinary disorders) | 3 | 3
Urinary retention (Renal and urinary disorders) | 4 | 4
Urinary tract obstruction (Renal and urinary disorders) | 1 | 2
Urinary tract pain (Renal and urinary disorders) | 1 | 2
Urinary urgency (Renal and urinary disorders) | 2 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0
Penile erosion (Reproductive system and breast disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthmatic episode (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bilaterial pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypercapnic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 1
Other (Skin and subcutaneous tissue disorders) | 2 | 0
"Poison ivy" per patient, dermatitis on left forearm (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulceration gluteal fold bilaterally (Skin and subcutaneous tissue disorders) | 0 | 1
Blotchy red spot forearm (Skin and subcutaneous tissue disorders) | 1 | 0
Boils-Four on right leg only (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema & swelling of abd incision (Skin and subcutaneous tissue disorders) | 1 | 0
Rash in groin (Skin and subcutaneous tissue disorders) | 0 | 1
Redness in hands and feet (Skin and subcutaneous tissue disorders) | 1 | 0
Basal skin cancer (removed from the nose) (Skin and subcutaneous tissue disorders) | 1 | 0
Open wound to left hip (Skin and subcutaneous tissue disorders) | 0 | 1
Sebaceous cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Squamous cell carcinoma of the face (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Bilateral Blepharoplasty (Surgical and medical procedures) | 1 | 0
Colostomy Reversal (Surgical and medical procedures) | 1 | 0
Tooth extractions (Surgical and medical procedures) | 0 | 1
Surgical resection of neck cancer (Surgical and medical procedures) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Hematoma (Vascular disorders) | 0 | 1
Hot flashes (Vascular disorders) | 1 | 10
Hypertension (Vascular disorders) | 20 | 23
Hypotension (Vascular disorders) | 1 | 0
Peripheral ischemia (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT01940276/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-03): https://cdn.clinicaltrials.gov/large-docs/76/NCT01940276/ICF_001.pdf